CLINICAL TRIAL: NCT00276770
Title: NCI-Sponsored Trial for the Evaluation of Safety and Preliminary Efficacy Using [F18] Fluorothymidine (FLT) As a Marker of Proliferation in Patients With Primary Brain Tumors
Brief Title: Positron Emission Tomography Using Fluorothymidine F 18 in Finding Recurrent Disease in Patients With Gliomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 27318; UW-6230; NCI-7223
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma; adult anaplastic ependymoma; adult anaplastic oligodendroglioma; adult diffuse astrocytoma; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma; adult ependymoma; adult oligodendroglioma; recurrent adult brain tumor; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Ependymoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Brain Neoplasms; Glioma | interventions — alovudine; Magnetic Resonance Spectroscopy

INTERVENTIONS:
Other: fluorine F 18 fluorothymidine
Procedure: positron emission tomography

SUMMARY:
RATIONALE: Diagnostic procedures, such as positron emission tomography using fluorothymidine F 18, may be effective in finding recurrent disease in patients with gliomas.

PURPOSE: This clinical trial is studying how well positron emission tomography using fluorothymidine F 18 works in finding recurrent disease in patients with gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of fluorothymidine F 18 for visual and dynamic brain tumor images in patients with glial neoplasms.
* Determine, preliminarily, the efficacy of this drug.

Secondary

* Compare, preliminarily, the efficacy of this drug to fludeoxyglucose F 18 in differentiating tumor recurrence from radiation necrosis.
* Determine the optimal time to image post injection of this drug.

OUTLINE: This is a pilot, nonrandomized study.

Patients receive fluorothymidine F 18 IV over 1 minute and then undergo positron emission tomography (PET) scanning of the brain over 2 hours.

After completion of the PET scan, patients are followed for at least 1 month.

PROJECTED ACCRUAL: A total of 12 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Radiological or established histological diagnosis of glioma

  * WHO grade 2-4 disease
* Presence of a new or enlarging enhancing lesion on gadolinium-enhanced MRI after prior radiotherapy

  * Differentiation of recurrent tumor from radiation necrosis is not possible
* No clinically significant signs of uncal herniation, including any of the following:

  * Acute pupillary enlargement
  * Rapidly developing (i.e., over hours) motor changes
  * Rapidly decreasing level of consciousness

PATIENT CHARACTERISTICS:

* Platelet count ≥ 75,000/mm^3
* WBC ≥ 3,000/mm^3
* Gamma-glutamyl-transferase ≤ 5 times upper limit of normal (ULN)
* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 10 g/dL
* SGOT and SGPT ≤ 2 times ULN
* Alkaline phosphatase ≤ 2 times ULN
* Lactic dehydrogenase ≤ 2 times ULN
* Direct and total bilirubin normal
* Amylase normal
* Haptoglobin normal
* Serum electrolytes normal
* CBC with platelets normal
* PT, PTT normal
* BUN and creatinine normal
* Not pregnant or lactating
* Urinalysis normal
* Negative pregnancy test
* Female patients must be postmenopausal for ≥ 1 year or surgically sterile, or on 1 of the following methods of birth control for ≥ 1 month: IUD, oral contraceptives, Depo-Provera, or Norplant

  * These criteria can be waived at the discretion of the investigator if the patient's intracranial tumor is considered life threatening and the 1-month wait required is not in the best interest of the patient
* No known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals
* No known HIV positivity
* Not requiring monitored anesthesia for positron emission tomography scanning

PRIOR CONCURRENT THERAPY:

* Concurrent biopsy or neurosurgical procedure for diagnostic and/or therapeutic purposes for this cancer allowed
* Concurrent surgery for this cancer allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-02; Primary Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander M. Spence, MD, Study Chair — University of Washington
Locations (1):
- University Cancer Center at University of Washington Medical Center, Seattle, Washington, United States

REFERENCES:
- [Result] Spence AM, Muzi M, Link JM, Hoffman JM, Eary JF, Krohn KA. NCI-sponsored trial for the evaluation of safety and preliminary efficacy of FLT as a marker of proliferation in patients with recurrent gliomas: safety studies. Mol Imaging Biol. 2008 Sep;10(5):271-80. doi: 10.1007/s11307-008-0151-6. Epub 2008 Jun 10. PMID 18543042